CLINICAL TRIAL: NCT01491958
Title: Phase II Trial Evaluating the Safety and Efficacy of Atorvastatin for the Prophylaxis of Acute Graft Versus Host Disease(GVHD) in Patients With Hematological Malignancies Undergoing HLA-Matched Related Donor Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Safety & Efficacy of Atorvastatin for Prophylaxis of Acute Graft Versus Host Disease in Patients With Hematological Malignancies HLA- Donor Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Yvonne Efebera, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-11004; NCI-2011-03590 (Registry Identifier: Clinical Trial Reporting Program (CTRP))
Record Dates: First submitted 2011-12-09; First posted 2011-12-14 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Acute Myelogenous Leukemia; Acute Lymphocytic Leukemia; Myelodysplastic Syndrome
Keywords: Leukemia; AML; ALL; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Leukemia | interventions — Atorvastatin; Tacrolimus; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Donor (Experimental): Related donors will receive atorvastatin 40 mg/day orally at least 14 days before anticipated first day of stem cell leukapheresis (LP) until successful completion of leukapheresis according to institutional guidelines. Peripheral blood stem cells will not be manipulated or T-depleted prior to administration.
  Interventions: Drug: atorvastatin
- Patient (Experimental): Patients will receive atorvastatin 40 mg starting at least 7 days before initiation of transplant conditioning regimen, to permit a 1 week observation period to rule out any atorvastatin-induced side effects before initiation of transplant conditioning. Patients will continue on atorvastatin with standard GVHD prophylaxis with tacrolimus and methotrexate until end of GVHD prophylaxis according to institutional standard guidelines, or until development of endpoint, which ever should occur first. Standard post transplant care will be administered.
  Interventions: Drug: atorvastatin; Drug: Tacrolimus; Drug: methotrexate

INTERVENTIONS:
Drug: atorvastatin — donors-will receive atorvastatin 40 mg/day orally at least 14 days before anticipated first day of stem cell leukapheresis (LP) until successful completion of leukapheresis according to institutional guidelines.
  Patients-will receive atorvastatin 40 mg starting at least 7 days before initiation of transplant conditioning regimen, to permit a 1 week observation period to rule out any atorvastatin-induced side effects before initiation of transplant conditioning. Patients will continue on atorvastatin with standard GVHD prophylaxis with tacrolimus and methotrexate until end of GVHD prophylaxis according to institutional standard guidelines, or until development of endpoint, which ever should occur first.
  Other Names: Lipitor
Drug: Tacrolimus — beginning on Day -2 through approximately Day +180 (that is, approximately 6 months after Day 0)
  Other Names: Prograf
  Arms: Patient
Drug: methotrexate — Day +1, +3, and +6 and +11
  Other Names: Amethopterin; MTX
  Arms: Patient

SUMMARY:
Phase II trial evaluating the safety & efficacy of Atorvastatin for prophylaxis of Acute Graft Versus Host Disease (GVHD) in patients with hematological malignances undergoing human leukocyte antigen (HLA)-Matched Related Donor Hematopoietic Stem Cell Transplant (HSCT).

DETAILED DESCRIPTION:
The study is a single-arm phase II single institutional trial evaluating the safety and efficacy of atorvastatin for the prophylaxis of acute GVHD in patients with hematological malignancies undergoing HLA matched related donor HSCT. This study will explore a two-pronged acute GVHD prophylaxis strategy, consisting of pre-treating consenting related donors with atorvastatin before stem cell mobilization and collection, followed by atorvastatin plus methotrexate/tacrolimus-based GVHD prophylaxis in transplant recipient patients.

ELIGIBILITY:
Inclusion Criteria:

Donor Eligibility Criteria

* The donor must be at least 18 years of age, and willing/able to provide informed consent. Complete medication list will be reviewed for potential negative interaction with atorvastatin.
* The donor must be an HLA-matched sibling or relative.
* Syngeneic donors are not eligible.
* Female donors of child-bearing potential should have a negative pregnancy test, and must not be breast feeding.
* Bilirubin, AST and ALT must be < 2 x normal; and absence of hepatic fibrosis/cirrhosis.
* Adequate renal function as defined by a serum creatinine clearance of ≥ 40% of normal calculated by Cockcroft-Gault equation.
* Adequate cardiac function with no history of congestive heart failure, uncontrolled atrial fibrillation or ventricular tachyarrhythmias.

Patient Eligibility Criteria

* Have hematologic malignancy requiring allogeneic HSCT, have adequate organ function, a serologic (or higher resolution) 6/6 class I human leukocyte antigen (HLA)-A and B and molecular class II DRB1 matched related donor, and are able to give informed consent.
* Patients > 18 and ≤ 65 years with comorbidity score ≤ 3 will be eligible for myeloablative conditioning (MAC), while patients > 65 years of age, those with previous history of autologous transplantation, or high comorbidity index (>3) will be eligible for reduced intensity conditioning (RIC) transplantation .
* All patients must have at least one 6/6 HLA-matched sibling donor.
* Patient must provide informed consent
* Patients must have left ventricular ejection fraction > 30%, no uncontrolled arrhythmias or New York Heart Association class III-IV heart failure.
* Bilirubin must be < 2 x normal; and absence of hepatic fibrosis/cirrhosis.
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) must be <2 x normal; and absence of hepatic fibrosis/cirrhosis.
* Serum creatinine clearance of ≥40% of normal calculated by Cockcroft-Gault equation.
* Forced expiratory volume in one second (FEV1)and diffusion capacity; corrected for hemoglobin(DLCO) ≥ 50% and 40% of predicted respectively.
* Karnofsky performance status > 70.
* A negative pregnancy test will be required for all women of child bearing potential. Breast feeding is not permitted.
* No HIV infection. Patients with immune dysfunction are at a significantly higher risk of toxicities from intensive immunosuppressive therapies.
* No evidence of active bacterial, viral or fungal infection at the time of transplant conditioning.
* No active alcohol or substance abuse within 6 months of study entry.
* Prior allogeneic transplant is acceptable.
* No history of intolerance or allergic reactions with atorvastatin or other statins.
* Patients who have previously been taking atorvastatin or any other statin will be eligible as long as there is no contraindication to switch to atorvastatin 40mg/day in the opinion of the treating physician.

Exclusion Criteria:

* Patients undergoing a T-cell depleted allogeneic transplantation will not be eligible.
* Patients receiving another investigational drug are not eligible unless cleared by Principal Investigator. Patients with prior malignancies except resected basal cell carcinoma, treated carcinoma in-situ, or other hematologic diseases for which allogeneic HSCT is a treatment strategy, are not eligible. Cancer treated with curative intent < 5 years previously will not be allowed unless approved by the Principal Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-12-10 (Actual); Primary Completion 2014-01-01 (Actual); Study Completion 2016-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Efebera, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who are candidates for HSCT using HLA matched related donors were eligible to be enrolled in the study.
Groups:
- Patients: Patients will receive atorvastatin 40 mg starting at least 7 days before initiation of transplant conditioning regimen, to permit a 1 week observation period to rule out any atorvastatin-induced side effects before initiation of transplant conditioning. Patients will continue on atorvastatin with standard GVHD prophylaxis with tacrolimus and methotrexate until end of GVHD prophylaxis according to institutional standard guidelines, or until development of endpoint, which ever should occur first. Standard post transplant care will be administered.
- Donors: Related donors will receive atorvastatin 40 mg/day orally at least 14 days before anticipated first day of stem cell leukapheresis (LP) until successful completion of leukapheresis according to institutional guidelines. Peripheral blood stem cells will not be manipulated or T-depleted prior to administration.
Period: Overall Study
Arm/Group | Patients | Donors
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients | Donor | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Median (Full Range); unit: years] | 51 [27 to 71] | 50 [25 to 68] | 51 [25 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 20 | 20 | 40
Region of Enrollment [Number; unit: patients]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Grades II to IV aGVHD at Day +100 of Atorvastatin Administration
Description: The incidence of grades II to IV aGVHD at day +100 of atorvastatin administration. The grading of aGVHD and cGVHD were done using the Consensus Conference criteria.
Time Frame: Up through day 100 following transplant
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Patients
Number analyzed (Participants) | 40
percentage of patients | 30 [17 to 45]

2. Secondary Outcome: Safety of Atorvastatin in Transplant Recipients in Terms of Adverse Events and Toxicities.
Description: Adverse events and toxicities were monitored in patients using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 criteria.
Time Frame: Patients: Baseline, weekly for 9 weeks and then on days 84, 91-100, 180 and 365. Donors: at apheresis and then 30 days later.
Population: Only patients with evaluable data reported
Measure: Number; unit: patients
Arm/Group | Patients
Number analyzed (Participants) | 36
patients
  Grade 2 elevated liver enzymes | 2
  Grade 4 elevated liver enzymes | 1

3. Secondary Outcome: Time to Neutrophil and Platelet Engraftment
Description: Neutrophil engraftment will be defined as first of three consecutive days with ANC ≥ 0.5 x 109/L post-conditioning regimen induced nadir. Similarly platelet engraftment is defined as first day of platelet count ≥ 20,000 x 109/L, without transfusion for 7 consecutive days.
Time Frame: weekly for 12 weeks, 100 days, 6 months, and 12 months
Measure: Median (Full Range); unit: days
Arm/Group | Patients
Number analyzed (Participants) | 40
days
  Neutrophil engraftment | 18 [13 to 26]
  Platelet engraftment | 14 [9 to 29]

4. Secondary Outcome: Percentage of Patients With Chronic Graft Versus Host Disease (cGVHD)
Description: cGVHD occurring anytime after day 100 post transplant will be termed chronic GVHD, and evaluated in patients who were followed for at least 100 days without early progression or death. Grading of cGVHD was done using the National Institutes of Health Consensus Development Project Criteria
Time Frame: up 1 year post transplant
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Patients
Number analyzed (Participants) | 34
percentage of patients | 43 [32 to 69]

5. Secondary Outcome: Non Relapse Mortality (NRM) at One Year
Description: Cumulative incidence of NRM will be calculated as the time from transplant until death not related to disease, where the competing risk for NRM was death due to disease. Patients who had not died were censored at last follow up.
Time Frame: up to 12 months post transplant
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Patients: Patients will receive atorvastatin 40 mg starting at least 7 days before initiation of transplant conditioning regimen, to permit a 1 week observation period to rule out any atorvastatin-induced side effects before initiation of transplant conditioning. Patients will continue on atorvastatin with standard GVHD prophylaxis with tacrolimus and methotrexate until end of GVHD prophylaxis according to institutional standard guidelines, or until development of endpoint, which ever should occur first. Standard post transplant care will be administered.
  atorvastatin: donors-will receive atorvastatin 40 mg/day orally at least 14 days before anticipated first day of stem cell leukapheresis (LP) until successful completion of leukapheresis according to institutional guidelines. Patients-will receive
Arm/Group | Patients
Number analyzed (Participants) | 40
percentage of patients | 5.5 [0.9 to 16.5]

ADVERSE EVENTS:
Description: Adverse events were assessed for 36 patients only using the Common Toxicity Criteria for Adverse Events version 4.0 (CTCAE v4.0)
Arm/Group | Patients
Serious Adverse Events (participants affected / at risk) | 5/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients (N=36)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Alanine Aminotransferase increased (Investigations) | 1 (1)
Aspartate Aminotransferase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients (N=36)
Anemia (Blood and lymphatic system disorders) | 14 (16)
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 (4)
Palpitations (Cardiac disorders) | 2 (2)
Sinus Tachycardia (Cardiac disorders) | 2 (2)
Endocrine Disorders (Endocrine disorders) | 2 (3)
Blurred Vision (Eye disorders) | 2 (2)
Dry eye (Eye disorders) | 4 (4)
Eye Disorders (Eye disorders) | 2 (3)
Abdominal Pain (Gastrointestinal disorders) | 6 (7)
Constipation (Gastrointestinal disorders) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 19 (26)
Dry mouth (Gastrointestinal disorders) | 9 (11)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 20 (21)
Nausea (Gastrointestinal disorders) | 24 (33)
Oral pain (Gastrointestinal disorders) | 4 (5)
Vomiting (Gastrointestinal disorders) | 10 (16)
Edema limbs (General disorders) | 7 (8)
Fatigue (General disorders) | 28 (34)
Fever (General disorders) | 10 (14)
General Disorder (General disorders) | 5 (6)
Localized Edema (General disorders) | 2 (3)
Pain (General disorders) | 11 (14)
Infections (Infections and infestations) | 15 (18)
Rhinitis Infective (Infections and infestations) | 2 (2)
Upper Respiratory Infection (Infections and infestations) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 8 (9)
Brusing (Injury, poisoning and procedural complications) | 2 (2)
Alanine Aminotransferase Increased (Investigations) | 26 (47)
Alkaline Phosphatase Increased (Investigations) | 12 (15)
Aspartate Aminotransferase Increased (Investigations) | 26 (49)
Blood Bilirubin Increased (Investigations) | 6 (6)
Cholesterol High (Investigations) | 4 (4)
Creatinine Increased (Investigations) | 25 (40)
INR Increased (Investigations) | 2 (2)
Investigations-other (Investigations) | 2 (2)
Lymphocyte Count Decreased (Investigations) | 2 (2)
Neutrophil Count Decreased (Investigations) | 9 (11)
Platelet Count Decreased (Investigations) | 12 (18)
Weight loss (Investigations) | 4 (4)
White Blood Cell Decreased (Investigations) | 10 (20)
Anorexia (Metabolism and nutrition disorders) | 13 (18)
Hypercalcemia (Metabolism and nutrition disorders) | 5 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 23 (35)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (3)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 18 (28)
Hypocalcemia (Metabolism and nutrition disorders) | 18 (32)
Hypokalemia (Metabolism and nutrition disorders) | 11 (12)
Hypomagnesemia (Metabolism and nutrition disorders) | 24 (50)
Hyponatremia (Metabolism and nutrition disorders) | 18 (33)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (4)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Muscleskeletal and Connective Tissues Disorder (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Dizziness (Nervous system disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 5 (6)
Headache (Nervous system disorders) | 9 (14)
Peripheral Sensory Neuropathy (Nervous system disorders) | 5 (7)
Anxiety (Psychiatric disorders) | 3 (3)
Confusion (Psychiatric disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 3 (3)
Acute Kidney Injury (Renal and urinary disorders) | 5 (5)
Chronic Kidney Disease (Renal and urinary disorders) | 2 (3)
Hematuria (Renal and urinary disorders) | 2 (2)
Renal and Urinary disorders (Renal and urinary disorders) | 5 (9)
Urinary Frequency (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 3 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (8)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 3 (4)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 13 (15)
Skin and subcutaneous tissue disorder (Skin and subcutaneous tissue disorders) | 3 (3)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 7 (7)
Hypotension (Vascular disorders) | 6 (6)
Thromboembolic event (Vascular disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No